CLINICAL TRIAL: NCT00974116
Title: MEND Childhood Obesity Treatment Programme: An RCT to Improve Body Composition and Cardiovascular Health in Overweight and Obese Children.
Brief Title: Trial of the MEND Childhood Obesity Treatment Program
Acronym: MEND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Child Health (Other)
Responsible Party: Professor Atul Singhal, Institute of Child Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08NT07
Record Dates: First submitted 2009-09-07; First posted 2009-09-10 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: MEND Childhood Obesity Program — The number of children who are obese in the UK is steadily increasing with both short and long term consequences for health. The aim of this study is to determine whether the MEND Programme (a new national initiative for the treatment of childhood obesity) is a successful and sustainable treatment for childhood obesity and obesity related health problems.
Behavioral: Control Group — No intervention

SUMMARY:
The number of children who are obese in the UK is steadily increasing with both short and long term consequences for health. The aim of this study is to determine whether the MEND Programme (a new national initiative for the treatment of childhood obesity) is a successful and sustainable treatment for childhood obesity and obesity related health problems.

300 overweight and obese children will be randomly assigned to start immediately on the MEND Programme for 6 months or join a waiting-list control group for 6 months. Measurements of health outcomes will be taken at baseline, and at 6, 12 and 24 months after the Programme. After 6 months of waiting-list time, the control group will follow the same protocol as the immediate starters. The researchers will be unaware (blinded) to which group each child has been assigned to. The study will examine the effects of the MEND Programme on body composition, cardiovascular health and psychological health.

DETAILED DESCRIPTION:
The Study is a Randomised Controlled Trial.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in the MEND Programme who are yet to be given a start date for the programme.
* Aged between 7-13 years old.
* Overweight or obese as defined by a BMI which falls above the 91st centile on the boys/girls BMI chart UK cross-sectional reference data:1997/1).
* Clinically well with no known chronic illness.

Exclusion Criteria:

* Age less than 7 years or older than 13.
* Known chronic illness.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index z-score | 6 months

SECONDARY OUTCOMES:
Body fat, waist circumference, blood pressure, arterial stiffness, heart rate control, fitness, physical activity and sedentary behaviour status, self esteem and health related quality of life. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof Atul Singhal, Principal Investigator — Institute of Child Health